CLINICAL TRIAL: NCT03683147
Title: RCT of Online Mindfulness-Based Stress Reduction for Metastatic Breast Cancer Patients
Brief Title: Mindfulness-Based Stress Reduction in Helping Participants With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 50317; NCI-2018-00453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 50317 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (online sessions, content manual, CD after 6 weeks) (Experimental): Participants randomized to the wait-list control condition complete the online intervention as in the intervention arm after the initial 6-week period has ended.
  Interventions: Other: Laboratory Biomarker Analysis; Behavioral: Meditation-Based Stress Reduction Program; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Intervention (online sessions, content manual, relaxation CD) (Experimental): Participants receive online group sessions over 60 minutes for 6 weeks, including 15 minutes of practice on that session's topic and daily meditation or yoga for 45 minutes. At the conclusion of the study period participants participate in mindfulness meditation over 3 hours. Participants also receive a content manual and relaxation CD.
  Interventions: Other: Laboratory Biomarker Analysis; Behavioral: Meditation-Based Stress Reduction Program; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Behavioral: Meditation-Based Stress Reduction Program — Participate in 6-week online program
  Other Names: MBSR; MBSR(BC); Meditation-Based Stress Reduction; Meditation-Based Stress Reduction (Breast Cancer); Meditation-Based Stress Reduction for Breast Cancer
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized trial studies how well a mindfulness-based stress reduction program helps participants with breast cancer that has spread to other places in the body. A cancer diagnosis is a life-changing and highly stressful event for most people, often resulting in marked declines in quality of life both during and after treatment. There are approximately 3 million women living with a history of invasive breast cancer in the U.S., with at least 150,000 living with metastatic disease. Patient preferences suggest a high need for complementary and alternative medicine interventions to address these chronic symptoms. Mindfulness-based stress reduction programs may help women living with metastatic breast cancer manage symptoms related to cancer treatment and improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a novel online mindfulness-based stress reduction (MBSR) treatment for distressed metastatic breast cancer patients in the hope of reaching patients otherwise unable to participate in traditional interventions due to high symptom burden.

II. Determine the impact of the intervention on both patient self-report and biological symptom measures.

OUTLINE: Participants are randomized to 1 of 2 arms.

INTERVENTION ARM: Participants receive online group sessions over 60 minutes for 6 weeks, including 15 minutes of practice on that session's topic and daily meditation or yoga for 45 minutes. At the conclusion of the study period participants participate in mindfulness meditation over 3 hours. Participants also receive a content manual and relaxation compact disc (CD).

CONTROL ARM: Participants randomized to the wait-list control condition complete the online intervention as in the intervention arm after the initial 6-week period has ended.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic breast cancer within the past 5 years and treated at Roswell Park Cancer Institute (RPCI)
* Ability to read and understand English
* Current distress score of 4+ on the National Comprehensive Cancer Network (NCCN) distress thermometer
* Access to an Internet connection with own device (computer, tablet, smartphone, etc.)
* Patient not currently involved in an ongoing psychological intervention
* If taking prescribed medication for mood or anxiety disorder, dosage has been consistent for prior 3 months

Exclusion Criteria:

* Unable to speak and understand English
* Prior or current experience with mindfulness-based practice
* Diagnosis of a psychotic disorder, bipolar disorder, substance abuse disorder, or reported suicidality
* Current involvement in any other psychological treatment (excluding medication) during study duration
* Currently being treated for another cancer diagnosis other than metastatic breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of the online intervention for metastatic breast cancer patients | At 6 weeks
  Successfully completing 4 out of 6 week sessions of online intervention for distressed metastatic breast cancer patients.

SECONDARY OUTCOMES:
Improvement in depression as measured by the Brief Symptom Inventory (BSI-18) | Baseline and 6 weeks
  BSI-18 - a self reported screening inventory to detect states of depression, anxiety and emotional distress.
Improvement in anxiety as measured by BSI-18 | Baseline and 6 weeks
  Self reported screening inventory designed to assess participants level of anxiety.
Improvement in fatigue measured with the Functional Assessment of Cancer Therapy Fatigue questionnaire | Baseline and 6 weeks
  Measured using the Functional Assessment of Cancer Therapy Fatigue (FACT-Fatigue). A questionnaire assessing fatigue.
Improvement in sleep impairment as measured by General Sleep Disturbance Scale | Baseline and 6 weeks
  Measured using the General Sleep Disturbance Scale - A 21 item scale rating specific sleep problems from 0 (not at all) to 7 (every day) used to evaluate sleep disturbance
Improvement in pain | Baseline and 6 weeks
  Visual analog scales will be used to assess multiple pain dimensions per the National Comprehensive Cancer Network (NCCN) guidelines for adult cancer pain.
Improvement in quality of life (QOL): FACT-B | Baseline 6 weeks
  This will be measured with the Functional Assessment of Cancer Comparisons made between the baseline and post-intervention assessment (6-week) will utilize one-sided permutation paired t-tests; with bootstrap or non-parametric methods considered as appropriate.
Improvement in blood pressure | Baseline and 6 weeks
  Blood pressure will be taken twice at each of the study time-points to ensure an accurate reading. All outcome measures are treated as quantitative variables and will be summarized by cohort and time-point using the appropriate descriptive statistics. Comparisons made between the baseline and post-intervention assessment (6-week) will utilize one-sided permutation paired t-tests; with bootstrap or non-parametric methods considered as appropriate.
Improvement in cancer-related biomarkers | Baseline and 6 weeks
  A panel of 25 cytokines reflecting Th1, Th2, and Th17 immunity will be collected, including (GMCSF, IFN-v, IL-1f3, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12, IL-13, IL-15, IL-17A, IL-17F, IL-17E/IL-25, IL-21, IL-22, IL-23, IL-27, IL-28A, IL-31, IL-33, MIP-3a/CCL20, TNFa, TNF|3). To visualize the pattern of immunologic markers that jointly distinguish intervention arms, hypothesis
Increases in mindfulness | Baseline and 6 weeks
  This will be measured with the Five Facet Mindfulness Questionnaire - (FFMQ). A questionnaire to explore mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chen Hong, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States